CLINICAL TRIAL: NCT01267084
Title: An Open-Label, Multicenter Study to Assess the Potential Effects of Ketoconazole on the Pharmacokinetics of Trabectedin in Subjects With Advanced Malignancies
Brief Title: A Study to Assess the Potential Effects of Ketoconazole on the Pharmacokinetics of Trabectedin in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017539; ET743OVC1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Neoplasm Metastases
Keywords: Trabectedin (YONDELIS); Ketoconazole; Antineoplastic Agents; Solid tumors; Locally advanced or metastatic disease; Chemotherapy; Pharmacokinetics
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Trabectedin; Ketoconazole; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part 1 (Experimental): Patients will receive trabectedin+ketoconazole followed by trabectedin alone. Each cycle will be will be separated by 21 days. Patients will receive 6 total consecutive doses of ketoconazole. Dexamethasone or equivalent steroid will be administered before trabectedin in each cycle.
  Interventions: Drug: Trabectedin; Drug: Ketoconazole; Drug: Dexamethasone or equivalent steroid
- Part 2 (Experimental): Patients will receive 1 of 2 treatment sequences; Sequence 1: trabectedin+ketoconazole followed by trabectedin alone or Sequence 2: trabectedin alone followed by trabectedin+ketoconazole. Each cycle will be separated by 21 days. Patients will receive 15 total consecutive doses of ketoconazole. Dexamethasone or equivalent steroid will be administered before trabectedin in each cycle.
  Interventions: Drug: Trabectedin; Drug: Ketoconazole; Drug: Dexamethasone or equivalent steroid

INTERVENTIONS:
Drug: Trabectedin — Patients will receive trabectedin 1.3 mg/m2 when given alone and 0.2mg/m2 when given with ketoconazole, intravenously (into a vein) for 3-hour.
Drug: Ketoconazole — Patients will receive ketoconazole 1 X 200 mg tablet, two times a day, orally (by mouth)
Drug: Dexamethasone or equivalent steroid — Patients will receive dexamethasone 20 mg or equivalent steroid intravenously, 30 minutes before trabectedin in each cycle.

SUMMARY:
The purpose of this study is to evaluate the potential effects of ketoconazole on blood levels of trabectedin after administration to patients with advanced malignancies.

DETAILED DESCRIPTION:
This is an open-label study (patients will know the names of the study drugs they receive), randomized (patients will be assigned 1 of 2 treatment sequences by chance) that is designed to examine the pharmacokinetics (blood levels) of trabectedin when coadministered with ketoconazole in patients with advanced malignancies. Study drugs include trabectedin and ketoconazole. Trabectedin is a drug being developed to treat patients with cancer that will be administered intravenously (IV) through a catheter (tube) into a central vein over a period of 3 hours once every 21 days with and without ketoconazole. Ketoconazole is an antifungal agent taken as tablets orally (by mouth), that may interfere with the metabolism of trabectedin. In addition, dexamethasone or equivalent steroid, a drug used to prevent nausea and vomiting in chemotherapy patients that may have protective effects on the liver, will be administered to patients before the administration of trabectedin in each treatment cycle. This study will consist of 2 parts, Part A and B. In Part A, trabectedin+ketoconazole followed by trabectedin alone will be administered with ketoconazole to 4 patients to evaluate safety. If the safety and PK data collected in Part A is deemed acceptable, enrollment in Part B of the study will begin and patients will receive 1 of 2 treatment sequences of trabectedin and ketoconazole. Patients in Part A and Part B who complete the treatment phase of the study or who are discontinued due to ketoconazole toxicity, and who in the opinion of the investigator would derive an overall clinical benefit from further treatment with trabectedin will have the opportunity to continue treatment with trabectedin in the optional extension phase. The dose and schedule of trabectedin may be modified by the treating physician in the optional extension phase to be more appropriate for the type of malignancy being treated. Patients will receive 20 mg of IV dexamethasone or equivalent steroid prior to trabectedin administration in all cycles. Part A consists of ketoconazole 200mg 2x daily+trabectedin 0.2mg/m2 i.v. followed 21 days later by trabectedin 1.3mg/m2 i.v. Part B consists of Sequence 1 (ketoconazole 200mg 2x daily+trabectedin 0.2mg/m2 i.v.followed 21 days later by trabectedin 1.3mg/m2 i.v.) and Sequence 2 (trabectedin 1.3mg/m2 i.v followed 21 days later by ketoconazole 200mg 2x daily+trabectedin 0.2mg/m2 i.v). Dexamethasone 20mg i.v. or equivalent, will be given 30 minutes before trabectedin in each cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic disease, any solid tumor except hepatocellular carcinoma (cancer of the liver), who have been relapsed or had progressive disease following standard of care treatment with chemotherapy prior to enrollment, or intolerant to prior standard of care treatment with chemotherapy

Exclusion Criteria:

* Patients with previous exposure to trabectedin
* Patients with cancer that has metastasized (spread) to the central nervous system
* Patients with known liver disease
* Patients who had a myocardial infarct (heart attack) within 6 months before enrollment or who have any other clinically significant or unstable medical condition as assessed by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of trabectedin | At protocol-specified time points for up to 8 days during each 21-day cycle in Sequence 1 and Sequence 2
Pharmacokinetics of ketoconazole | 1 day during Sequence 1 or Sequence 2 after ketoconazole is coadministered with trabectedin
  This will be measured when ketoconazole will be administered.

SECONDARY OUTCOMES:
Number of patients with adverse events | Time from 1st dose of trabectedin up to 30 days after the last dose of trabectedin
Findings from clinical laboratory evaluations | Time from 1st dose of trabectedin up to 30 days after the last dose of trabectedin
Findings from vital signs measurements | Time from 1st dose of trabectedin up to 30 days after the last dose of trabectedin
Findings from physical examinations | Time from 1st dose of trabectedin up to 30 days after the last dose of trabectedin
Evaluation of Survival data | At a time point to be determined by the sponsor at a later date

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- Belgium (2):
  - Brussels
  - Wilrijk

REFERENCES:
- [Derived] Machiels JP, Staddon A, Herremans C, Keung C, Bernard A, Phelps C, Khokhar NZ, Knoblauch R, Parekh TV, Dirix L, Sharma S. Impact of cytochrome P450 3A4 inducer and inhibitor on the pharmacokinetics of trabectedin in patients with advanced malignancies: open-label, multicenter studies. Cancer Chemother Pharmacol. 2014 Oct;74(4):729-37. doi: 10.1007/s00280-014-2554-1. Epub 2014 Aug 7. PMID 25100135
- See also: An Open-Label, Multicenter Study to Assess the Potential Effects of Ketoconazole on the Pharmacokinetics of Trabectedin in Subjects with Advanced Malignancies — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=871&filename=CR017539_CSR.pdf